CLINICAL TRIAL: NCT02088437
Title: High Intensity Physiotherapy for Hip Fractures in the Acute Hospital Setting
Brief Title: High Intensity Physiotherapy for Hip Fractures
Acronym: HIP4hips
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Alfred (Other)
Responsible Party: Principal Investigator, Lara Kimmel, Principal Investigator, The Alfred
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 32/14
Record Dates: First submitted 2014-03-06; First posted 2014-03-17 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (Active Comparator): usual care physiotherapy - once daily treatment whilst inpatient in acute hospital
  Interventions: Other: Usual Care
- Intensive physiotherapy (Experimental): additional once daily physiotherapy and once daily allied health assistant intervention
  Interventions: Other: Intensive physiotherapy

INTERVENTIONS:
Other: Intensive physiotherapy — additional once daily physiotherapy and once daily allied health assistant intervention (equals two more treatments) whilst an inpatient in acute hospital
  Arms: Intensive physiotherapy
Other: Usual Care — once daily physiotherapy whilst acute hospital inpatient
  Arms: Usual care

SUMMARY:
Every day, more than 40 Australian break their hip, Most are over the age of sixty five. Hip fractures are a significant problem for the older people, the hospital system and community as a whole because of the increasing numbers of fractures and the cost of hospitalisation and ongoing care. After one year, less than half of all people with a hip fracture can walk as well as they did before the fracture. Physiotherapy in the acute hospital setting is an integral part of patient care, although the intensity of physiotherapy a patient receives is variable and the optimal number of treatment sessions per day remains unknown. Studies in other patient groups have shown that increased physiotherapy can improve patient outcomes by increasing muscle strength and mobility. It can also reduce the negative effects of bed rest such as muscle wasting, blood clots in the lungs or leg veins and chest infections such as pneumonia. This study aims to investigate the effectiveness of an intensive physiotherapy program in hip fracture patients to further understand this and the effect it has on patient function.

In this research the investigators will randomly allocate patients into 2 groups; usual care and intensive physiotherapy. The usual care group will have physiotherapy treatment daily whereas the intensive physiotherapy group will have an additional daily treatment by a physiotherapist as well as a daily treatment by an allied health assistant. The objectives are to achieve better functional outcomes in the patient's hospital stay (ie improved mobility), reduce the time for patients to be physically ready to go home, increase the number of patients able to go directly home or to fast stream rehabilitation (rather than a slow stream option).

If increased intensity of physiotherapy is found to improve patient's mobility outcomes, this research will provide the confidence to endorse a change to current clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Admission to The Alfred with an isolated hip fracture and treated with internal fixation, aged 65 or above

Exclusion Criteria:

* fracture is in the sub-trochanteric region of the femur,
* if it is pathological,
* if post operative orders are for non-weight bearing on the operated hip,
* if they were unable to mobilise independently (or with gait aid) prior to admission,
* or if they were admitted from a nursing home.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 92 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
modified IOWA Level of Assistance Scale | 5 days
  Functional score measuring 6 mobility domains

SECONDARY OUTCOMES:
length of stay - acute and rehabilitation | participants will be followed for duration of hospital stay - average one month
  the length of acute hospital stay and rehabilitation stay - until discharge home or to a long term facility
timed up and go | 5 days
Glasgow Outcomes Score -Extended | 6 months
discharge destination | participants will be followed until discharge from the acute hospital - average 10 days
  discharge destination from the acute hospital - options include: home, fast stream rehabilitation, slow stream rehabilitation, long term facility
physical readiness for discharge | average one month
  when a patient is deemed physically ready go home - eg can access their house and mobilise within house and outdoors
12-Item Short Form Health Survey (SF-12) | 6 months
EuroQOL five dimensions questionnaire (EQ-5D) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lara A Kimmel, B.Physio, Principal Investigator — The Alfred
Locations (1):
- The Alfred, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Kimmel LA, Liew SM, Sayer JM, Holland AE. HIP4Hips (High Intensity Physiotherapy for Hip fractures in the acute hospital setting): a randomised controlled trial. Med J Aust. 2016 Jul 18;205(2):73-8. doi: 10.5694/mja16.00091. PMID 27456448